CLINICAL TRIAL: NCT02400892
Title: Patent Foramen Ovale and the Risk of Postoperative Delirium Following Elective Hip and Knee Arthroplasty Surgeries
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Daniel Bainbridge, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 105952
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Foramen Ovale, Patent; Delirium; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Foramen Ovale, Patent; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PFO: Subjects with a bedside Transthoracic Echocardiogram (TTE) bubble study positive for a PFO
  Interventions: Other: TTE Bubble Study
- Control: Subjects with a bedside TTE bubble study negative for a PFO
  Interventions: Other: TTE Bubble Study

INTERVENTIONS:
Other: TTE Bubble Study — Bedside transthoracic echocardiogram bubble study to assess for the presence or absence of a PFO

SUMMARY:
This study will involve patients who are planned to have hip or knee replacement surgeries. They will undergo a Transthoracic Echocardiogram study (an ultrasound of the heart) to look for a Patent Foramen Ovale (PFO). A PFO is a hole in the heart that everyone is born with and in most cases eventually closes by adulthood. However, it does not always close in all people. The investigators will compare the participants as two groups - those with a PFO, and those without, and look for differences in delirium in their postoperative stay. This will help us look for an association between postoperative delirium and the presence of a PFO.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo an elective, primary hip replacement surgery or knee replacement surgery
* Fluent in English

Exclusion Criteria:

* Planned to undergo a revision knee or hip replacement
* History of cardiac surgery or prosthetic heart valves
* History of other structural heart abnormalities, not involving the atrial septum
* History of preexisting neurologic condition that affects the patient's day-to-day life, including a history of Dementia, Stroke, or previous Neurosurgery causing ongoing problems
* Significant visual problems felt by investigators to impair Confusion Assessment Method use
* Significant hearing problems felt by investigators to impair Confusion Assessment Method use
* History of psychiatric problems requiring treatment with major antidepressant drugs or antipsychotic drugs
* History of a Deep Venous Thrombosis or Pulmonary Embolism in the past year
* History of known Atrial Fibrillation in the past 3 months
* Presence of a pacemaker or implantable cardioverter-defibrillator
* History of Transient Ischemic Attack or Stroke within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will involve adult patients planned to undergo an elective, primary hip or knee replacement surgery at one of the hospitals of the London Health Sciences Centre (University Hospital or Victoria Hospital).
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium - measured by Confusion Assessment Method (CAM) Scores positive for delirium | Daily CAM assessment starting Postoperative Day #1 after surgery until discharge or up to 1 week postoperatively

SECONDARY OUTCOMES:
Length of hospital stay | Postoperative length of hospital stay after surgery( expected mean of 4 days)
Major adverse events (including Heart Attack, Stroke, Heart failure, Blood clots, Abnormal heart rhythms, other major complications, and death) | Postoperative period until hospital discharge (expected mean of 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bainbridge, MD, FRCPC, Principal Investigator — Western University
Locations (1):
- University Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Gai N, Lavi R, Jones PM, Lee H, Naudie D, Bainbridge D. The use of point-of-care ultrasound to diagnose patent foramen ovale in elective hip and knee arthroplasty patients and its association with postoperative delirium. Can J Anaesth. 2018 Jun;65(6):619-626. doi: 10.1007/s12630-018-1073-7. Epub 2018 Jan 24. PMID 29368313